CLINICAL TRIAL: NCT00573755
Title: Phase II Randomized Study of Sorafenib Compared to Placebo When Administered in Combination With Aromatase Inhibitors for Postmenopausal Women With Metastatic Breast Cancer
Brief Title: Sorafenib and Letrozole, Anastrozole, or Exemestane in Treating Postmenopausal Women With Estrogen Receptor-Positive and/or Progesterone Receptor-Positive Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of participant accrual
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC0731; P30CA015083 (NIH); RC0731 (Other: Mayo Clinic Cancer Center); 07-005768 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral sorafenib tosylate twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: letrozole; Drug: sorafenib tosylate
- Arm II (Active Comparator): Patients receive oral placebo twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: anastrozole; Drug: exemestane; Drug: letrozole; Other: placebo

INTERVENTIONS:
Drug: anastrozole — given orally
Drug: exemestane — given orally
Drug: letrozole — given orally
Drug: sorafenib tosylate — given orally
  Arms: Arm I
Other: placebo — given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Aromatase inhibition therapy using letrozole, anastrozole, or exemestane may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether sorafenib is more effective than a placebo when given together with letrozole, anastrozole, or exemestane in treating metastatic breast cancer.

PURPOSE: This randomized phase II trial is studying how well sorafenib works compared with a placebo when given together with letrozole, anastrozole, or exemestane in treating postmenopausal women with estrogen receptor-positive and/or progesterone receptor-positive metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the progression-free survival of postmenopausal women with estrogen receptor- and/or progesterone receptor-positive metastatic breast cancer treated with sorafenib tosylate vs placebo and letrozole, anastrozole, or exemestane.

Secondary

* To compare the overall survival and time to treatment failure of patients treated with these regimens.
* To compare the objective tumor response rate and duration of response in patients treated with these regimens.
* To assess the adverse event profile of sorafenib tosylate in combination with aromatase inhibitors in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior aromatase inhibitor therapy (yes vs no) and line of endocrine therapy for metastatic disease (first-line vs second-line). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral sorafenib tosylate twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28.
* Arm II: Patients receive oral placebo twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (i.e., MRI or CT scan of chest, abdomen and pelvis) or ≥ 10 mm by spiral CT scan

  * Non-measurable disease allowed, defined as all other lesions (or sites of disease), including small lesions (longest diameter < 20 mm by conventional techniques or < 10 mm by spiral CT scan)
* Must have objective evidence of progression within the past 3 months
* No human epidermal growth factor receptor 2 (HER2)/neu overexpression, defined as gene amplification by fluorescence in situ hybridization or 3+ overexpression by immunohistochemistry, or unknown HER2/neu status
* No active brain metastases

  * Patients with neurological symptoms must undergo a contrast CT scan or MRI of the brain to exclude active brain metastasis
  * Patients with treated brain metastases allowed provided they have no evidence of disease and have been off definitive therapy (including steroids) for the past 3 months
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive disease

PATIENT CHARACTERISTICS:

* Female
* The Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Postmenopausal
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* INR ≤ 1.5
* PTT within normal limits
* Creatinine ≤ 1.5 times ULN
* Not nursing, pregnant, or able to become pregnant
* No significant traumatic injury within the past 4 weeks
* No history of bleeding diathesis or uncontrolled coagulopathy
* No serious, nonhealing wound, ulcer, or bone fracture
* No clinically significant cardiac disease, including any of the following:

  * New York Heart Association class III-IV congestive heart failure
  * Unstable angina (i.e., anginal symptoms at rest) or new-onset angina (i.e., began within the past 3 months)
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring antiarrhythmic therapy
* No uncontrolled hypertension (systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg), despite optimal medical management
* No thrombolic, embolic, venous, or arterial events (e.g., cerebrovascular accident including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage or bleeding event > grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ grade 3 within the past 4 weeks
* No active clinically serious infection > grade 2
* No known HIV infection
* No chronic hepatitis B or C infection
* No previous or concurrent cancer that is distinct in primary site or histology from breast cancer except carcinoma in situ of the cervix, treated basal cell skin cancer, superficial bladder tumors (i.e., Ta and Tis), or any cancer curatively treated within the past 5 years
* No known or suspected allergy to sorafenib tosylate or other agents used in this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No major surgery or open biopsy within the past 4 weeks
* No more than 1 prior regimen of endocrine therapy for metastatic breast cancer, provided that the patient has not received an aromatase inhibitor within the past 12 months
* No more than 1 prior regimen of chemotherapy for metastatic disease
* More than 2 weeks since prior radiotherapy, except if to a non-target lesion only or single-dose radiotherapy for palliation

  * Prior radiotherapy to a target lesion(s) is permitted only if there has been clear progression of the lesion since radiotherapy was completed
* Concurrent anticoagulation treatment (e.g., warfarin or heparin) allowed
* No concurrent Hypericum perforatum (St. John's wort), rifampin, bevacizumab, or any other drugs (licensed or investigational) that target vascular endothelial growth factor (VEGF) or VEGF receptors
* No concurrent cytochrome P450 enzyme-inducing anti-epileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Roy, MD, Study Chair — Mayo Clinic; Donald W Northfelt, M.D., Principal Investigator — Mayo Clinic; Timothy J Hobday, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four (4) participants were recruited at Mayo Clinic between January 2008 and August 2008. This trial was terminated early due to lack of participant accrual.
Groups:
- Sorafenib Plus Aromatase Inhibitor: Patients receive oral sorafenib tosylate twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
- Placebo Plus Aromatase Inhibitor: Patients receive oral placebo twice daily and oral letrozole, anastrozole, or exemestane once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Still receiving treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.9) | 54.5 (4.9) | 61.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the earliest date of documentation of disease progression or death due to any cause. In the case of a participant started treatment and then never return for any evaluations, the participant was censored for progression 1 day post-randomization.
Time Frame: Time from randomization to disease progression or death (up to 5 years)
Population: All participants who have met the eligibility criteria, signed a consent form and were randomized to one of the two treatment groups were evaluable for the primary endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 2 | 2
months | NA [NA to NA] — There is not enough events reported to compute median and 95% Confidence Interval (CI). | NA [NA to NA] — One participant had a progression at 12.5 months. There is not enough events reported to compute median and 95% CI.

2. Secondary Outcome: Overall Survival
Description: Survival time was defined as the time from randomization to death due to any cause.
Time Frame: Time from randomization to death (up to 5 years)
Population: The number of patients enrolled in the study does not allow for meaningful analysis for this outcome. All patients were alive at the time of their last treatment follow up.
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from the date of the randomization to the date at which the patient was removed from treatment due to progression, adverse events, or refusal.
Time Frame: Time from randomization to treatment failure (up to 5 years)
Population: The number of patients enrolled in the study does not allow for meaningful analysis for this outcome.
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Objective Tumor Response Rate
Description: A confirm response was defined as either a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluation at least 4 weeks apart. The confirmed response rate was estimated within each treatment group by the number of confirmed responses divided by the total number of participants randomized.
Time Frame: Up to 5 years
Population: The number of patients enrolled in the study does not allow for meaningful analysis for this outcome.
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response was defined for all patients who have achieved a confirmed response as the date at which the patient's earliest best objective status was first noted to be either a CR or PR to the earliest date progression was documented.
Time Frame: Up to 5 years
Population: The number of patients enrolled in the study does not allow for meaningful analysis for this outcome.
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Event
Description: Number of participants that experienced adverse events (grade 3 and above) as measured by NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Adverse events were assessed every week during first 6 weeks of therapy, every 4 weeks on months 1 to 6, every 12 weeks on months 7 and beyond and at the end of treatment.
Time Frame: Time from randomization to end of treatment
Measure: Number; unit: participants
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Number analyzed (Participants) | 2 | 2
participants
  Fatigue | 1 | 0
  Hemoglobin decreased | 1 | 0
  Mucositis oral | 1 | 0
  Muscle weakness | 1 | 0
  Platelet count decreased | 1 | 0
  Serum potassium increased | 1 | 0
  Thrombotic microangiopathy | 1 | 0
  Serum sodium decreased | 1 | 0
  Mucositis oral (clin exam) | 1 | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib Plus Aromatase Inhibitor | Placebo Plus Aromatase Inhibitor
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Plus Aromatase Inhibitor (N=2) | Placebo Plus Aromatase Inhibitor (N=2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib Plus Aromatase Inhibitor (N=2) | Placebo Plus Aromatase Inhibitor (N=2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1) | 1 (6)
Hypothyroidism (Endocrine disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 0 (0)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (17) | 1 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight loss (Investigations) | 1 (1) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (21) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (2)
Hypertension (Vascular disorders) | 1 (10) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes